CLINICAL TRIAL: NCT04951024
Title: Comparison of Perioperative Analgesia Effectiveness Between Thoracolumbal Interfascial Plane Block With Erector Spinae Plane Block In Lumbar Posterior Decompression and Stabilization: A Study to Interleukin-6 and Interleukin-10 Plasma Concentration, Pain Scale, Total Opioid Consumption, and Cardiovascular Stability
Brief Title: Thoracolumbal Interfascial Plane Block Versus Erector Spinae Plane Block for Lumbar Posterior Decompression Stabilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes105
Record Dates: First submitted 2021-06-26; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Lumbar Posterior Decompression
Keywords: Thoracolumbal Interfascial Plane Block; Erector Spinae Plane Block; Lumbar Posterior Decompression and Stabilization
MeSH Terms: interventions — Dental Occlusion; Parapsychology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracolumbar interfacial plane (TLIP) Block (Experimental): Thoracolumbar interfacial plane (TLIP) Block will be performed after induction of anesthesia by anesthesiologist who is not part of investigators for this study. Bilateral 20 ml 0.25 % Bupivacaine injected between multifidus and longissimus muscle with Ultrasound guidance.
  Interventions: Procedure: Thoracolumbar interfacial plane (TLIP) Block; Procedure: Erector Spinae Plane (ESP) Block
- Erector Spinae Plane (ESP) Block (Active Comparator): Erector Spinae Plane (ESP) Block will be performed after induction of anesthesia by anesthesiologist who is not part of investigators for this study. Bilateral 20 ml 0.25 % Bupivacaine injected between the erector spinae muscles and transverse process with Ultrasound guidance
  Interventions: Procedure: Thoracolumbar interfacial plane (TLIP) Block; Procedure: Erector Spinae Plane (ESP) Block

INTERVENTIONS:
Procedure: Thoracolumbar interfacial plane (TLIP) Block — TLIP Block: Bilateral 20 ml 0.25 % Bupivacaine injected between multifidus and longissimus muscle with Ultrasound guidance.
Procedure: Erector Spinae Plane (ESP) Block — ESP Block: Bilateral 20 ml 0.25 % Bupivacaine injected between the erector spinae muscles and transverse process with Ultrasound guidance.

SUMMARY:
This study aimed to found out The Comparison Of Perioperative Analgesia Effectiveness Between Thoracolumbal Interfascial Plane Block with Erector Spinae Plane Block In Lumbar Posterior Decompression and Stabilization.

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial. Forty subject will be recruited with non-probability consecutive sampling method. Subjects who meet all inclusion criteria and do not have exclusion criteria will be asked to sign the informed consent form before included in this study. Subjects will be randomized into two groups. The first group is the group who will get Bilateral Thoracolumbal Interfascial Plane Block after general anesthesia and the second group will be the group who will get Bilateral Erector Spinae Plane Block after general anesthesia. After surgery, pain scale, time to first morphine dose, total morphine consumption in 24 hours, cardiovascular stability and adverse events will be recorded for both group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years old
2. Patients schedule for elective posterior decompression and stabilization lumbar spine surgery
3. ASA I - III
4. Decompression and posterior stabilization's patients who didn't caused by infection or abscess

Exclusion Criteria:

1. Patients who refuse to participate in this study
2. Body Mass Index < 18,5 kg/m2 and > 27,0 kg/m2
3. Patient with history of chronic opioid
4. Patient with coagulation disorder
5. Patient with cognitive disorders
6. Infection at the injection area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Interleukin-6 and Interleukin-10 at 6 hours after Lumbar Posterior Decompression and Stabilization | Before surgery and 6 hours after surgery
  Measure by ELISA

SECONDARY OUTCOMES:
investigators will record total morphine dose needed in 24 hours | 24 hours after surgery
  investigators will record time to first morphine dose after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tantri AR, Rahmi R, Marsaban AHM, Satoto D, Rahyussalim AJ, Sukmono RB. Comparison of postoperative IL-6 and IL-10 levels following Erector Spinae Plane Block (ESPB) and classical Thoracolumbar Interfascial Plane (TLIP) block in a posterior lumbar decompression and stabilization procedure: a randomized controlled trial. BMC Anesthesiol. 2023 Jan 10;23(1):13. doi: 10.1186/s12871-023-01973-w. PMID 36624374